CLINICAL TRIAL: NCT02679521
Title: The Effectiveness of Extracorporeal Shock Wave Therapy for Patients With Plantar Fasciitis Who Satisfy a Clinical Prediction Rule
Brief Title: Radial Extracorporeal Shock Wave Treatment for Chronic Plantar Fasciopathy
Acronym: RSWT_CPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr Mahmoud Ibrahim Ibrahim (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr Mahmoud Ibrahim Ibrahim, Scientist, Rocky Mountain University of Health Professions
Organization: Rocky Mountain University of Health Professions (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 070609-02
Record Dates: First submitted 2016-02-03; First posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Fasciitis, Plantar
Keywords: Extracorporeal Shock Wave Therapy; Painful Heel; Plantar fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rESWT (Active Comparator): Radial extracorporeal shock wave therapy (rESWT).
  Interventions: Device: ESWT
- Placebo (Placebo Comparator): Placebo treatment.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: ESWT — Radial extracorporeal shock wave therapy (rESWT) was performed by the principal investigator with a Swiss DolorClast device (EMS Electro Medical Systems Corporation; Dallas, Texas, USA).
  The Swiss DolorClast device obtained Pre-Market Approval (PMA) by FDA as Class III orthopedic lithotripsy device to treat heel pain associated with chronic proximal plantar fasciitis on May 8, 2007 (PMA # P050004), and was re-classified as Class III Generator, Shock Wave, For Pain Relief (Product Code NBN) in the Spring 2009. The present study started on October 3, 2007.
  Each patient received two sessions of rESWT one week apart, with 2,000 impulses per session (air pressure of the device set at 3.5 bar; impulses applied with the 15 mm applicator at frequency of 8 Hz).
  Other Names: Swiss DolorClast
  Arms: rESWT
Device: Placebo — Placebo treatment was performed identically as rESWT but with a clasp on the heel that prevented transmission of the impulses from the applicator to the skin at the treatment site.
  Arms: Placebo

SUMMARY:
Radial extracorporeal shock wave therapy (rESWT) has been previously demonstrated as an efficient treatment option for heel pain associated with chronic proximal plantar fasciitis when administered in three sessions. The present study tested the hypothesis that heel pain associated with chronic proximal plantar fasciitis can also be treated successfully with rESWT when only two treatment sessions are performed.

DETAILED DESCRIPTION:
Plantar fasciitis, the most common cause of heel pain, accounts for approximately 11-15% of foot symptoms presenting to physicians. In the United States, more than two million individuals are treated for PF on an annual basis. The term Plantar Fasciitis implies an inflammatory condition by the suffix 'itis'. However, various lines of evidence indicate that this disorder is better classified as 'fasciosis' or 'fasciopathy'. Details about etiology, pathogenesis, risk factors, diagnosis and general treatment strategies for plantar fasciitis have been provided in a series of comprehensive reviews recently. Briefly, both athletes and the elderly commonly present to physicians with plantar fasciitis, and the diagnosis of plantar fasciitis is usually based on the patient's history and clinical examination. It has been recommended in the literature to start treatment of plantar fasciitis with conservative treatment modalities, including physical therapy, stretching, inserts/orthotics etc. For patients not responding to conservative treatment for 6 months (between 10% and 20% of all patients) extracorporeal shock wave therapy (ESWT) should be considered. In case a patient does not benefit from ESWT either, surgical intervention should be taken into account.

Several randomized, controlled trials of ESWT with focused shock waves for chronic plantar fasciitis were published, demonstrating favourable results in the range of 50% to 70% after a followup period of three months after treatment. Besides this, a recent study demonstrated safety and efficacy of radial extracorporeal shock wave therapy (rESWT) for chronic plantar fasciitis (Gerdesmeyer et al., Am J Sports Med 2008 Nov;36(11):2100-9). These authors administered rESWT or placebo treatment in three sessions, each two weeks (±4 days) apart and evaluated the treatment outcome at twelve weeks and twelve months after the first session. The authors found a statistically significant (p < 0.05) difference in the reduction of the mean Visual Analog Scale composite score between the patients treated with rESWT and the placebo-treated patients both at twelve weeks and twelve months from baseline.

To further evaluate the potential of rESWT to become a routine therapeutic modality in the treatment of chronic plantar fasciitis, the investigators of the present study identified the following questions not addressed in the study by Gerdesmeyer et al. (2008). First, it is unknown whether treatment success can also be reached by two rESWT sessions one week apart, rather than by three rESWT sessions each two weeks apart as applied by Gerdesmeyer et al. (2008). Anecdotal reports by colleagues in Europe indicated that this could indeed be the case. Second, immediate return to normal daily life activities (including sports activities) and normal daily shoe wear indicates that patients suffering from chronic plantar fasciitis and treated with rESWT experience profound pain relief already much earlier than three months after the first rESWT session, applied as first followup in the study by Gerdesmeyer et al. (2008).

Therefore the hypothesis was tested in the present prospective, randomized, double-blinded, placebo-controlled study that treatment of chronic plantar fasciopathy with two rESWT sessions one week apart will result in profound pain relief compared to placebo treatment already four weeks after the first rESWT treatment, lasting for at least six months.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 years
* Diagnosis of painful heel syndrome by clinical examination, with the following positive clinical signs: (i) pain in the morning or after sitting a long time; (ii) local pain where the fascia attaches to the heel; and (iii) increasing pain with extended walking or standing for more than 15 minutes
* History of six months of unsuccessful conservative treatment
* Therapy free period of at least four weeks before referral
* Signed informed consent

Exclusion Criteria:

* Bilateral plantar fasciitis
* Dysfunction of foot or ankle (for example, instability)
* Arthrosis or arthritis of the foot
* Infections or tumors of the lower extremity
* Neurological abnormalities, nerve entrapment (for example, tarsal tunnel syndrome)
* Vascular abnormality (for example, severe varicosities, chronic ischemia)
* Operative treatments of the heel spur
* Hemorrhagic disorders and anticoagulant therapy
* Pregnancy
* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pain (VAS score) | Change from Baseline Pain Score (VAS) at 6 months.

SECONDARY OUTCOMES:
Quality of life (modified Roles & Maudsley score) | Change from Baseline Quality of Life Score (R&M) at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud I Ibrahim, PhD, PT, Principal Investigator — Rocky Mountain University of Health Professions, Provo, UT 84601, USA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ibrahim MI, Donatelli RA, Schmitz C, Hellman MA, Buxbaum F. Chronic plantar fasciitis treated with two sessions of radial extracorporeal shock wave therapy. Foot Ankle Int. 2010 May;31(5):391-7. doi: 10.3113/FAI.2010.0391. PMID 20460065